CLINICAL TRIAL: NCT05422833
Title: Effectiveness of Medical Management in the Field of Rare Diseases. The Example of Fibrous Dysplasia of Bone.
Brief Title: Effectiveness of Medical Management of Fibrous Dysplasia of Bone.
Acronym: Efficience
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 370
Record Dates: First submitted 2022-05-10; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Fibrous Dysplasia of Bone; McCune Albright Syndrome
Keywords: Fibrous Dysplasia of Bone; McCune Albright Syndrome; rare; bone disease; healthcare organization
MeSH Terms: conditions — Fibrous Dysplasia of Bone; Fibrous Dysplasia, Polyostotic; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before: Children and adults with FD/MAS who visited at least once in our center (outpatient and hospitalized patients).
  and with the first visit in the center included between 1996 and 2006 - before certification of our center.
  Interventions: Other: Evaluation and analysis of clinical data
- After: Children and adults with FD/MAS who visited at least once in our center (outpatient and hospitalized patients).
  and with the first visit in the center included between 2007 and 2019 - after certification of our center.
  Interventions: Other: Evaluation and analysis of clinical data

INTERVENTIONS:
Other: Evaluation and analysis of clinical data — Evaluation and analysis of clinical data (baseline demographic features (sex, age at diagnosis, age at first symptoms, age at first visit), initial presenting symptoms, affected bone sites (monostotic FD or polyostotic FD), renal phosphate wasting, MAS, Mazabraud syndrome, endocrine disease, fractures, bone specific treatment especially bisphosphonate and surgery, pain and disease's severity.

SUMMARY:
The objective of our study was to assess the effectiveness of our reference center since its constitution.

In a retrospective cohort study, we compared the activity of our center, including the time elapsed between diagnosis and access to the center and the diagnostic delay of patients with fibrous dysplasia between two periods, 1996-2006 (before certification of our center) and 2007-2019 (after certification of our center).

ELIGIBILITY:
Inclusion Criteria:

We have included children and adults with FD/MAS who visited at least once in our center (outpatient and hospitalized patients). The diagnosis was established by an expert of the center, based on clinical, biological, imaging and/or histological arguments

Exclusion Criteria:

The absence of detectable bone lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with FD/MAS who visited at least once in our center
Sampling Method: Non-Probability Sample
Enrollment: 528 (Actual)
Dates: Start 1996-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
to compare time elapsed between first symptomes or discovery of bone lesions and the diagnosis of FD | 1996-2019
  The main objective was to compare time elapsed between first symptomes or discovery of bone lesions and the diagnosis of FD, over 2 periods of time: 1996-2006 (before certification) and 2007-2019 (after certification).

CONTACTS AND LOCATIONS:
Locations (1):
- rheumatology department, hopital Edouard Herriot, Lyon, France